CLINICAL TRIAL: NCT00460538
Title: Efficacy and Safety of Lectranal® in Treatment of Seasonal Allergic Rhinitis Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milsing d.o.o. (Other)
Responsible Party: Neven Tudoric MD PhD, Dubrava University Hospital, Zagreb, Croatia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIL-002
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Last update posted 2010-04-05 (Estimated); Status verified 2010-03

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Seasonal allergic rhinitis; lectranal; allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: placebo
- 1 (Active Comparator)
  Interventions: Dietary Supplement: Lectranal

INTERVENTIONS:
Dietary Supplement: Lectranal — Dosage form: capsule
  1: Dosage: 2 capsule Frequency and duration: 2 times daily over the 6 weeks
  Arms: 1
Dietary Supplement: placebo — Dosage form: capsule 2: Dosage: 2 capsules Frequency and duration: 2 times daily over the 6 weeks
  Arms: 2

SUMMARY:
The purpose of the study is to determine weather Lectranal is effective in treatment of seasonal allergic rhinitis symptoms.

DETAILED DESCRIPTION:
Patients allergic to the specific pollen are divided into two groups randomly. One group is being administered Lectranal and the other group is being administered placebo during the period of 6 weeks in season of the pollen. Methods used for evaluation are: SARS questionnaire(seasonal allergic rhinitis symptoms), Mini RQLQ (mini rhinoconjunctivitis quality of life questionnaire) skin Prick test, specific IgE and IgG, eosinophilia in nasal secretion. Methods used for follow up safety include side effects report, physical examination and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* history of seasonal allergic rhinitis symptoms to pollen
* positive skin prick test to pollen
* negative history of seasonal allergic asthma
* male or female older than 18
* female participants must use appropriate contraception
* able to comply to study procedures

Exclusion Criteria:

* pregnancy
* alcohol or drug abuse
* subject receiving antihistamines , immunotherapy or on hyposensibilisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
changes in SARS (seasonal allergic rhinitis symptoms) | 6 weeks
changes in Mini RQLQ (mini rhinoconjunctivitis quality of life questionnaire) | 6 weeks
changes in specific IgE | 6 weeks
changes in specific IgG | 6 weeks

SECONDARY OUTCOMES:
Prick test change | 6 weeks
change in eosinophilia in nasal secretion | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neven Tudoric, MD PhD, Principal Investigator — Dubrava University Hospital
Locations (1):
- Dubrava University Hospital, Zagreb, Croatia

REFERENCES:
- [Result] Matkovic Z, Zivkovic V, Korica M, Plavec D, Pecanic S, Tudoric N. Efficacy and safety of Astragalus membranaceus in the treatment of patients with seasonal allergic rhinitis. Phytother Res. 2010 Feb;24(2):175-81. doi: 10.1002/ptr.2877. PMID 19504468